CLINICAL TRIAL: NCT03454607
Title: Safety and Feasibility Study of the Foot Controlled Robotic Endoscope Enabled Robot (FREE) in Functional Endoscopic Sinus Surgery
Brief Title: Foot Controlled Robotic Endoscope Enabled Robot FESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in patient recruitment
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jason Chan, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRE-2017.307-T
Record Dates: First submitted 2017-12-27; First posted 2018-03-06 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Sinusitis; Polyp of Nasal Sinus
Keywords: FREE; Robotic
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FREE robot (Experimental): Patients undergoing sinus surgery with the FREE robot
  Interventions: Device: FREE robot

INTERVENTIONS:
Device: FREE robot — FREE robot to hold endoscope

SUMMARY:
To evaluate the safety and feasibility of a Foot Controlled Robotic Endoscope Enabled Robot (FREE) in performing functional endoscopic sinus surgery to answer the two key questions:

1. Is the FREE robot feasible to use in patients for endoscopic sinus surgery?
2. Is the FREE robot safe to use in patients for endoscopic sinus surgery?

DETAILED DESCRIPTION:
Through previous cadaver experiments we have demonstrated and experimentally validated a new foot-controlled robotic endoscope holder prototype that allows the surgeon to directly manipulate surgical instruments with both hands at all times. The conducted ex-vivo cadaver test, corroborated the feasibility of the robotic prototype. However the next step requires further clinical trials to evaluate its use in endoscopic sinus surgery in patients that is the purpose of this study

ELIGIBILITY:
Inclusion Criteria:

* Undergoing FESS surgery for benign pathology

Exclusion Criteria:

* Pregnant/ lactating female patients
* Younger than 18 years of age
* Cognitive impairment or unable to provide informed consent
* Malignant sinus pathologies
* Previous endoscopic sinus surgery
* Contraindication to general anaesthesia
* Untreated active infection
* Non-correctable coagulopathy
* Emergency Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Conversion | Intraoperative
  The rate of conversions to normal holding of the endoscope
Perioperative complications | Within 30 days postoperative
  Assessment of perioperative complications

SECONDARY OUTCOMES:
Surgical outcomes | Intraoperative and postoperative 2 weeks and 30 days
  Operative time
Surgical outcomes | Intraoperative and postoperative 2 weeks and 30 days
  Estimated blood loss
Surgical Outcomes | Intraoperative and postoperative 2 weeks and 30 days
  Length of stay
Quality of life | Within 30 days postoperative
  The Total Nasal Symptom Score (TNSS; possible score of 0-12) is the sum of 4 individual participant-assessed symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe. Higher scores represent a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No